CLINICAL TRIAL: NCT00510484
Title: A Double-blind, Randomized, Multi-center, Placebo-controlled, Cross-over Study to Assess the Efficacy and Safety of Pancrelipase Delayed Release 24,000 Unit Capsules in Subjects With Pancreatic Exocrine Insufficiency Due to Cystic Fibrosis
Brief Title: Study Investigating a Delayed-Release Pancrelipase in Patients With Exocrine Pancreatic Insufficiency Due to Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Djenane Bennett, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S245.3.126; 2007-004005-10
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Results first posted 2009-07-20 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2009-08

CONDITIONS: Cystic Fibrosis
Keywords: Pancreatic exocrine insufficiency; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Pancrelipase Delayed Release
- B (Placebo Comparator)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Pancrelipase Delayed Release — 24000 unit Capsule
  Arms: A
Drug: Placebo Comparator — Placebo
  Arms: B

SUMMARY:
This study will assess the effect of pancrelipase delayed release 24,000 unit capsules on fat and nitrogen absorption in subjects with PEI due to Cystic Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed CF diagnosis by two positive chloride sweat tests or gene analysis
* Confirmed PEI by historical CFA < 70% without supplementation or current or historical fecal elastase < 50µg/g stool (within the last 12 months)
* Subjects of 12 years or older
* Currently receiving treatment with a commercially available pancreatic enzyme product on a stable dose for more than 3 months
* Clinically stable condition without evidence of acute respiratory disease or any other acute condition
* Females of child-bearing potential must agree to continue using a medically acceptable method of birth control

Exclusion Criteria:

* Ileus or acute abdomen
* History of fibrosing colonopathy
* History of distal ileal obstruction syndrome within 6 months of enrollment
* Use of an immunosuppressive drug
* Any type of malignancy involving the digestive tract in the last 5 years
* Known infection with HIV

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (23):
- United States (19):
  - Site 11, Long Beach, California
  - Site 10, Los Angeles, California
  - Site 13, San Francisco, California
  - Site 5, Miami, Florida
  - Site 4, Orlando, Florida
  - Site 1, Iowa City, Iowa
  - Site 7, Louisville, Kentucky
  - Site 17, Boston, Massachusetts
  - Site 8, Ann Arbor, Michigan
  - Site 6, Minneapolis, Minnesota
  - Site 18, Long Branch, New Jersey
  - Site 16, Albuquerque, New Mexico
  - Site 19, Cincinnati, Ohio
  - Site 12, Dayton, Ohio
  - Site 2, Toledo, Ohio
  - Site 14, Oklahoma City, Oklahoma
  - Site 3, Hershey, Pennsylvania
  - Site 15, Philadelphia, Pennsylvania
  - Site 9, Nashville, Tennessee
- Site 20, Petrofi, Hungary
- Site 21, Jerusalem, Israel
- Site 22, Johannesburg, South Africa
- Site 23, Barcelona, Spain

REFERENCES:
- [Result] Trapnell BC, Maguiness K, Graff GR, Boyd D, Beckmann K, Caras S. Efficacy and safety of Creon 24,000 in subjects with exocrine pancreatic insufficiency due to cystic fibrosis. J Cyst Fibros. 2009 Dec;8(6):370-7. doi: 10.1016/j.jcf.2009.08.008. Epub 2009 Oct 7. PMID 19815466

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in 10 centers in US between November 2007 and January 2008. Before the randomization, subjects were evaluated for eligibility. They underwent a short period of up to 14 days on their usual pancreatic enzyme supplementation. Subjects were to take 4000 lipase units/g fat intake during both cross-over periods.
Pre-assignment Details: Two subjects prematurely withdrew before the randomization (1 withdrew consent and 1 for protocol violation). 32 subjects were randomly allocated to pancrelipase/placebo or placebo/pancrelipase. 1 subject did not complete the second period of the treatment. 1 subject was randomized twice and only the second randomization was used for analyses.
Period: Period 1
Arm/Group | Placebo/Pancrelipase | Pancrelipase/Placebo
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Wash-out Period
Arm/Group | Placebo/Pancrelipase | Pancrelipase/Placebo
Started | 16 | 16
Completed | 16 | 15
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Period 2
Arm/Group | Placebo/Pancrelipase | Pancrelipase/Placebo
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Pancrelipase | Pancrelipase/Placebo | Total
Number analyzed (Participants) | 16 | 16 | 32
Age Continuous [Mean (Standard Deviation); unit: years] | 22.2 (7.8) | 22.8 (6.5) | 22.5 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 12 | 9 | 21
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Coefficient of Fat Absorption (%)
Description: This coefficient is calculated from fat intake and fat excretion : 100*[fat intake-fat excretion]/fat intake. Stools were collected on 3 days during the 5 days treatment period. Higher values indicate a better response.
Time Frame: 5 days
Population: The analysis was done on the Full Analysis Sample defined as the randomized subjects with at least one post-baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Pancrelipase | Placebo
Number analyzed (Participants) | 31 | 31
Percentage | 88.62 (6.62) | 49.78 (18.33)
Statistical Analysis 1: Comparison: Pancrelipase vs Placebo; The parameter was analyzed using an analysis of variance (ANOVA) including treatment, sequence and period as fixed effect and subject within sequence as a random effect; Test type: Superiority or Other; p < 0.001, ANOVA

2. Secondary Outcome: Coefficient of Nitrogen Absorption (%)
Description: This coefficient is calculated from nitrogen intake and nitrogen excretion : 100*[nitrogen intake-nitrogen excretion]/nitrogen intake. Stools were collected on 3 days during the 5 days treatment period. Higher values indicate a better response.
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Pancrelipase | Placebo
Number analyzed (Participants) | 31 | 31
Percentage | 85.06 (6.38) | 49.99 (17.14)
Statistical Analysis 1: Comparison: Pancrelipase vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA

3. Secondary Outcome: Total Fat Excretion (Grams)
Description: Total amount of fat excreted during the stool collection period. Stools were collected on 3 days during the 5 days treatment period. Lower values indicate a better response.
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Pancrelipase | Placebo
Number analyzed (Participants) | 31 | 31
Grams | 57.7 (46.1) | 243.2 (112.7)
Statistical Analysis 1: Comparison: Pancrelipase vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA

4. Secondary Outcome: Total Stool Weight (Grams)
Description: Total weight of the stools collected during the stool collection period. Stools were collected on 3 days during the 5 days treatment period. Lower values indicate a better response.
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Pancrelipase | Placebo
Number analyzed (Participants) | 31 | 31
Grams | 630.1 (306.9) | 1582.5 (664.5)
Statistical Analysis 1: Comparison: Pancrelipase vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA

5. Secondary Outcome: Stool Frequency
Description: Stool frequency is the average of the daily number of stools recorded during the treatment period. Lower values indicate a better response.
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number per day
Arm/Group | Pancrelipase | Placebo
Number analyzed (Participants) | 32 | 31
Number per day | 1.75 (0.81) | 2.88 (1.18)
Statistical Analysis 1: Comparison: Pancrelipase vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA

6. Other Pre Specified Outcome: Percentage of Days With Formed/Normal Stools.
Description: The percentage of days with formed/normal stools is calculated from the diary during the treatment period: 100*(number of days with formed/normal stools/number of days with any stool). Higher values indicate a better response.
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Pancrelipase | Placebo
Number analyzed (Participants) | 32 | 31
Percentage of days | 75.0 (30.0) | 23.9 (27.8)
Statistical Analysis 1: Comparison: Pancrelipase vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA

7. Secondary Outcome: Percentage of Days With no Flatulence.
Description: The percentage of days with no flatulence is calculated from the diary during the treatment period: 100*(number of days with no flatulence/number of days recorded in diary). Higher values indicate a better response.
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Pancrelipase | Placebo
Number analyzed (Participants) | 32 | 31
Percentage of days | 41.6 (41.9) | 23.1 (35.1)
Statistical Analysis 1: Comparison: Pancrelipase vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.013, ANOVA

8. Secondary Outcome: Percentage of Days With no Abdominal Pain.
Description: The percentage of days with no abdominal pain is calculated from the diary during the treatment period: 100*(number of days with no abdominal pain / number of days recorded in diary). Higher values indicate a better response.
Time Frame: 5 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Pancrelipase | Placebo
Number analyzed (Participants) | 32 | 31
Percentage of days | 90.3 (16.8) | 59.1 (43.2)
Statistical Analysis 1: Comparison: Pancrelipase vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA

ADVERSE EVENTS:
Arm/Group | Pancrelipase | Placebo
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 14/32 | 20/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pancrelipase (N=32) | Placebo (N=31)
Faeces abnormal (Gastrointestinal disorders) | 1 | 6
Flatulence, Bloating and Distension (Gastrointestinal disorders) | 3 | 8
Gastrointestinal and abdominal pain (Excl oral and throat) (Gastrointestinal disorders) | 3 | 10
Physical Examination Procedures (Investigations) | 1 | 2
Headaches NEC (Nervous system disorders) | 2 | 7
Neurological signs and symptoms NEC (Nervous system disorders) | 2 | 0
Coughing and Associated Symptoms (Respiratory, thoracic and mediastinal disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Only treatment emergent events have been presented. They are defined as events started at or after the 1st administration of study medication and include events started prior to the 1st administration but which worsened after the 1st intake.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At 60 days prior to submitting or presenting a manuscript or other materials relating to the Study to a publisher, reviewer, or other outside persons, the Site shall provide to Sponsor a copy and allow Sponsor 60 days to review and comment.